CLINICAL TRIAL: NCT00565448
Title: International Randomized Study to Evaluate the Addition of Docetaxel to the Combination of Cisplatin-5-fluorouracil (TCF) vs. Cisplatin-5-fluorouracil (CF) in the Induction Treatment of Nasopharyngeal Carcinoma (NPC) in Children and Adolescents
Brief Title: Docetaxel in Combination With Cisplatin-5-fluorouracil for the Induction Treatment of Nasopharyngeal Carcinoma in Children and Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC10339; 2007-001211-33 (EudraCT Number)
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Results first posted 2010-03-25 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Nasopharyngeal Neoplasms; Carcinoma
Keywords: Nasopharyngeal carcinoma
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Carcinoma; Nasopharyngeal Carcinoma | interventions — Docetaxel; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Docetaxel/Cisplatin/5-FU (TCF) (Experimental): * Docetaxel 75 milligrams per square meter (mg/m²) over 1 hour on Day 1 every 3 weeks
  * Cisplatin 75 mg/m² Day 1 over 6 hours every 3 weeks
  * 5-Fluorouracil 750 mg/m²/day continuous infusion Days 1 to 4 every 3 weeks as an induction therapy
  Consolidation treatment: radiation therapy for 7-8 weeks and 3 cycles of cisplatin 100 mg/m² every 3 weeks.
  Interventions: Drug: docetaxel; Drug: cisplatin; Drug: 5-fluorouracil
- Cisplatin/5-FU (CF) (Active Comparator): * Cisplatin 80 mg/m² Day 1 over 6 hours every 3 weeks
  * 5-Fluorouracil 1000 mg/m²/day continuous infusion Day 1 to 4 every 3 weeks as an induction therapy.
  Consolidation treatment: radiation therapy for 7-8 weeks and 3 cycles of cisplatin 100 mg/m² every 3 weeks.
  Interventions: Drug: cisplatin; Drug: 5-fluorouracil

INTERVENTIONS:
Drug: docetaxel — Pharmaceutical form:solution for infusion
  Route of administration:intravenous
  Other Names: Taxotere®; XRP6976
  Arms: Docetaxel/Cisplatin/5-FU (TCF)
Drug: cisplatin — Pharmaceutical form:solution for infusion
  Route of administration:intravenous
Drug: 5-fluorouracil — Pharmaceutical form:solution for infusion
  Route of administration:intravenous
  Other Names: 5-FU

SUMMARY:
The primary objective is to estimate the Complete Response rate of docetaxel to the combination of cisplatin-5-fluorouracil (TCF) compared to cisplatin-5-fluorouracil (CF) in the Induction treatment of Nasopharyngeal Carcinoma (NPC).

The secondary objectives are to determine:

* the safety of TCF in comparison to CF after induction treatment of NPC,
* the pharmacokinetics of docetaxel when added to CF,
* the Overall Response rate of TCF and CF on completion of induction and consolidation (chemo-radiotherapy) treatment of NPC, and to compare overall survival between TCF and CF.

DETAILED DESCRIPTION:
Planned treatment duration:

* induction period: 9 weeks of induction treatment
* consolidation period: 9 weeks of chemoradiation treatment.

The consolidation treatment was the same for all participants: radiation therapy for 7-8 weeks and 3 cycles of cisplatin 100 mg/m² every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of nasopharyngeal carcinoma World Health Organization (WHO) type II or III
* Children and adolescents newly diagnosed with Stage IIB-IV NPC with measurable disease, who are >1 month to ≤21 years of age at the time of diagnosis. In France, participants must be ≥1 year to ≤21 years of age at the time of diagnosis

Exclusion Criteria:

* Participants with short life expectancy
* Prior chemotherapy or radiotherapy to the nasopharynx or neck for the treatment of nasopharyngeal carcinoma
* Inadequate renal function evidenced by unacceptable laboratory results

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2007-11; Primary Completion 2009-03 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (26):
- Investigational Site Number 012001, Algiers, Algeria
- Brazil (2):
  - Investigational Site Number 076002, Rio de Janeiro
  - Investigational Site Number 076001, São Paulo
- Investigational Site Number 156005, Fuzhou, China
- Investigational Site Number 250001, Villejuif, France
- India (4):
  - Investigational Site Number 356003, Ahmedabad
  - Investigational Site Number 356004, Kolkata
  - Investigational Site Number 356002, Thiruvananthapuram
  - Investigational Site Number 356001, Vellore
- Investigational Site Number 360001, Jakarta, Indonesia
- Investigational Site Number 380001, Milan, Italy
- Investigational Site Number 484001, Villahermosa, Mexico
- Morocco (3):
  - Investigational Site Number 504001, Casablanca
  - Investigational Site Number 504002, Rabat
  - Investigational Site Number 504003, Rabat
- Investigational Site Number 608002, Quezon City, Philippines
- South Korea (3):
  - Investigational Site Number 410001, Seoul
  - Investigational Site Number 410003, Seoul
  - Investigational Site Number 410002, Seoul
- Thailand (2):
  - Investigational Site Number 764001, Bangkok
  - Investigational Site Number 764002, Chiang Mai
- Tunisia (2):
  - Investigational Site Number 788002, Sousse
  - Investigational Site Number 788003, Tunis
- Turkey (Türkiye) (3):
  - Investigational Site Number 792003, Abacıoğlu
  - Investigational Site Number 792001, Ankara
  - Investigational Site Number 792002, Istanbul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from November 2007 until October 2008. The study was conducted at 26 centers in 14 countries.
Groups:
- Docetaxel /Cisplatin/5-FU: Docetaxel 75 mg/m² in combination with Cisplatin 75 mg/m² on Day 1 and 5-Fluorouracil 750 mg/m²/day on Days 1 to 4 every 3 weeks as induction therapy.
  Consolidation treatment: radiation therapy for 7-8 weeks and 3 cycles of cisplatin 100 mg/m² every 3 weeks.
- Cisplatin/5-FU: Cisplatin 80 mg/m² on Day 1 and 5-Fluorouracil 1000 mg/m²/day Days 1 to 4 every 3 weeks as induction therapy.
  Consolidation treatment: radiation therapy for 7-8 weeks and 3 cycles of cisplatin 100 mg/m² every 3 weeks.
Period: Overall Study
Arm/Group | Docetaxel /Cisplatin/5-FU | Cisplatin/5-FU
Started | 50 (Intent to treat (ITT) population: all randomized participants. All were treated.) | 25 (ITT population: all randomized participants. All were treated.)
Completed | 47 (Completed induction period as per protocol.) | 23 (Completed induction period as per protocol.)
Not Completed | 3 | 2
Not completed — Adverse Event | 1 | 2
Not completed — Disease progression | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT population: all randomized participants.
Groups:
- Cisplatin/5-FU: Cisplatin 80 mg/m² on Day 1 and 5-Fluorouracil 1000 mg/m²/day on Days 1 to 4 every 3 weeks as induction therapy.
  Consolidation treatment: radiation therapy for 7-8 weeks and 3 cycles of cisplatin 100 mg/m² every 3 weeks.
- Total: Total of all reporting groups
Arm/Group | Docetaxel /Cisplatin/5-FU | Cisplatin/5-FU | Total
Number analyzed (Participants) | 50 | 25 | 75
Age, Continuous [Median (Full Range); unit: years] | 16 [9 to 21] | 16 [9 to 21] | 16 [9 to 21]
Age, Customized [Number; unit: participants]
  Infants from 28 days to 23 months | 0 | 0 | 0
  Children from 2 years to <12 years | 4 | 1 | 5
  Adolescents from 12 years to <16 years | 20 | 10 | 30
  Adolescents >=16 | 26 | 14 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 6 | 21
  Male | 35 | 19 | 54

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response (CR)
Description: CR assessed by independent reviewers, according to the Modified Response Evaluation Criteria in Solid Tumors (RECIST) from the National Cancer Institute (NCI). Disease response evaluated after the completion of the induction treatment and prior to the radiation treatment. CR defined as the complete disappearance of the target and non-target lesion(s) identified at baseline after radiological evaluation by Magnetic Resonance Imaging (MRI) only.
Time Frame: after the completion of the induction treatment (up to 9 weeks)
Population: ITT population: all randomized participants.
Measure: Number; unit: participants
Groups:
- Docetaxel /Cisplatin/5-FU: Docetaxel 75 mg/m² in combination with Cisplatin 75 mg/m² on Day 1 and 5-Fluorouracil 750 mg/m²/day on Days 1 to 4 every 3 weeks as induction therapy
- Cisplatin/5-FU: Cisplatin 80 mg/m² on Day 1 and 5-Fluorouracil 1000 mg/m²/day on Days 1 to 4 every 3 weeks as induction therapy
Arm/Group | Docetaxel /Cisplatin/5-FU | Cisplatin/5-FU
Number analyzed (Participants) | 50 | 25
participants | 1 | 0
Statistical Analysis 1: Comparison: Docetaxel /Cisplatin/5-FU vs Cisplatin/5-FU; There was no formal power calculation. A selection design was used to determine how many participants would be accrued to correctly select the treatment group with the best CR rate with 80% probability; Test type: Superiority or Other; p = 1.0000, Fisher Exact — The Fisher's exact test was used to compare the CR proportions

2. Secondary Outcome: Docetaxel Area Under the Plasma Concentration-time Curve (AUC) in the Docetaxel/Cisplatin/5-FU Group
Description: AUC estimated by Bayesian method using concentration-time data for each participant and the previously defined adult population model as prior information (with validity of the estimation verified).
Time Frame: Three plasma samples: one just before then 45 minutes and 5hour after the end of cycle 1 infusion
Population: Participants who were randomized to docetaxel/cisplatin/5-FU and had evaluable docetaxel pharmacokinetic (PK) sample.
Measure: Mean (Standard Deviation); unit: µg*h/mL
Groups:
- Docetaxel/Cisplatin/5-FU: Docetaxel 75 mg/m² in combination with Cisplatin 75 mg/m² on Day 1 and 5-Fluorouracil 750 mg/m²/day on Days 1 to 4 every 3 weeks as induction therapy
Arm/Group | Docetaxel/Cisplatin/5-FU
Number analyzed (Participants) | 26
µg*h/mL | 3.43 (2.05)

3. Secondary Outcome: Overall Response (OR)
Description: OR is classified as CR, partial response (PR), stable disease (SD), progressive disease (PD) or Unknown on completion of both induction and radiation treatment and assessed according to the Modified RECIST from the NCI. CR is defined as the disappearance of all target lesions (TLs) and non-TLs. PR is defined as ≥30% decrease in the sum of the longest diameters (LD) of TLs, taking as reference the disease measurement done at study entry. PD is defined as ≥20% increase in the sum of the LD of TLs, taking as a reference the smallest disease measurement recorded at study entry or the appearance of ≥1 new lesions or unequivocal progression of non-TLs. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: after the completion of the consolidation treatment (up to 18 weeks)
Population: ITT population: all randomized participants.
Measure: Number; unit: participants
Groups:
- Docetaxel /Cisplatin/5-FU: Docetaxel 75 mg/m² in combination with Cisplatin 75 mg/m² on Day 1 and 5-Fluorouracil 750 mg/m²/day on Days 1 to 4 every 3 weeks as induction therapy.
  Consolidation Treatment: Radiation for 6 weeks and 3 cycles of platinum 100 mg/m² every 3 weeks.
- Cisplatin/5-FU: Cisplatin 80 mg/m² on Day 1 and 5-Fluorouracil 1000 mg/m²/day on Days 1 to 4 every 3 weeks as induction therapy.
  Consolidation Treatment: Radiation for 6 weeks and 3 cycles of platinum 100 mg/m² every 3 weeks.
Arm/Group | Docetaxel /Cisplatin/5-FU | Cisplatin/5-FU
Number analyzed (Participants) | 50 | 25
participants
  CR | 1 | 1
  PR | 43 | 20
  SD | 2 | 1
  PD | 2 | 0
  Unknown | 0 | 0
  Missing | 2 | 3

4. Secondary Outcome: Overall Survival (OS) Rate
Description: OS rate is the percentage of participants who survived 3 years after completion of consolidation treatment period. The Kaplan-Meier method was used to estimate OS rate.
Time Frame: 3 years after the end of the consolidation treatment period (up to 40 months from randomization)
Population: ITT population: all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Docetaxel /Cisplatin/5-FU | Cisplatin/5-FU
Number analyzed (Participants) | 50 | 25
percentage of participants | 85.7 [75.9 to 95.5] | 78.0 [60.8 to 95.1]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit regardless of seriousness or relationship to investigational product.
Description: Reported AEs are treatment-emergent AEs that is AEs that developed/worsened during the 'on treatment period' (from first dose up 30 days after administration of the last cycle [maximum 3 cycle]). Safety population: all subjects who received at least one cycle of any component of the study drug combination.
Arm/Group | Cisplatin/5-FU | Docetaxel /Cisplatin/5-FU
Serious Adverse Events (participants affected / at risk) | 11/25 | 20/50
Other Adverse Events (participants affected / at risk) | 23/25 | 49/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin/5-FU (N=25) | Docetaxel /Cisplatin/5-FU (N=50)
BONE MARROW FAILURE (Blood and lymphatic system disorders) | 1 | 0
FEBRILE BONE MARROW APLASIA (Blood and lymphatic system disorders) | 1 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 5
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 0
NEUTROPENIA/NEUTROPHIL COUNT (Blood and lymphatic system disorders) | 2 | 4
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 3
GASTRITIS (Gastrointestinal disorders) | 0 | 1
MALLORY-WEISS SYNDROME (Gastrointestinal disorders) | 0 | 1
PROCTALGIA (Gastrointestinal disorders) | 0 | 1
STOMATITIS (Gastrointestinal disorders) | 1 | 2
VOMITING (Gastrointestinal disorders) | 0 | 2
ASTHENIA (General disorders) | 0 | 1
PYREXIA (General disorders) | 1 | 2
HYPERSENSITIVITY (Immune system disorders) | 0 | 1
CENTRAL LINE INFECTION (Infections and infestations) | 1 | 0
NEUTROPENIC INFECTION (Infections and infestations) | 1 | 0
PHARYNGITIS BACTERIAL (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 1
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 | 1
SEPTIC SHOCK (Infections and infestations) | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1
BLOOD CREATININE INCREASED (Investigations) | 0 | 1
HAEMOGLOBIN DECREASED (Investigations) | 0 | 1
ANOREXIA (Metabolism and nutrition disorders) | 0 | 3
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 | 0
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
ATAXIA (Nervous system disorders) | 1 | 0
CONVULSION (Nervous system disorders) | 2 | 1
HEADACHE (Nervous system disorders) | 1 | 0
ACUTE PRERENAL FAILURE (Renal and urinary disorders) | 1 | 0
HYPOTENSION (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin/5-FU (N=25) | Docetaxel /Cisplatin/5-FU (N=50)
ANAEMIA (Blood and lymphatic system disorders) | 3 | 14
BONE MARROW FAILURE (Blood and lymphatic system disorders) | 1 | 3
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 6
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 | 6
NEUTROPENIA/NEUTROPHIL COUNT (Blood and lymphatic system disorders) | 7 | 20
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 3
OTOTOXICITY (Ear and labyrinth disorders) | 6 | 7
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 | 10
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 | 11
CONSTIPATION (Gastrointestinal disorders) | 0 | 7
DIARRHOEA (Gastrointestinal disorders) | 3 | 15
DRY MOUTH (Gastrointestinal disorders) | 5 | 9
DYSPEPSIA (Gastrointestinal disorders) | 0 | 3
DYSPHAGIA (Gastrointestinal disorders) | 7 | 12
NAUSEA (Gastrointestinal disorders) | 10 | 33
ODYNOPHAGIA (Gastrointestinal disorders) | 1 | 3
SALIVARY HYPERSECRETION (Gastrointestinal disorders) | 0 | 3
STOMATITIS (Gastrointestinal disorders) | 5 | 30
VOMITING (Gastrointestinal disorders) | 21 | 47
ASTHENIA (General disorders) | 0 | 5
FATIGUE (General disorders) | 1 | 8
MUCOSAL INFLAMMATION (General disorders) | 3 | 5
PYREXIA (General disorders) | 5 | 11
HYPERSENSITIVITY (Immune system disorders) | 0 | 4
FOLLICULITIS (Infections and infestations) | 0 | 5
ORAL CANDIDIASIS (Infections and infestations) | 0 | 8
SINUSITIS (Infections and infestations) | 3 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 3
OVERDOSE (Injury, poisoning and procedural complications) | 2 | 2
RADIATION SKIN INJURY (Injury, poisoning and procedural complications) | 1 | 11
THERMAL BURN (Injury, poisoning and procedural complications) | 2 | 5
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 3
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 4
PLATELET COUNT DECREASED (Investigations) | 0 | 3
WEIGHT DECREASED (Investigations) | 8 | 20
WEIGHT INCREASED (Investigations) | 1 | 4
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 2 | 7
ANOREXIA (Metabolism and nutrition disorders) | 5 | 21
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 | 4
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 6
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 6
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 6
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 | 0
DYSGEUSIA (Nervous system disorders) | 0 | 4
HEADACHE (Nervous system disorders) | 1 | 8
ANXIETY (Psychiatric disorders) | 0 | 4
DEPRESSION (Psychiatric disorders) | 0 | 3
NEPHROPATHY TOXIC (Renal and urinary disorders) | 0 | 4
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 5
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 8
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 4
PHARYNGEAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 4 | 3
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 | 29
DERMATITIS (Skin and subcutaneous tissue disorders) | 4 | 7
RASH (Skin and subcutaneous tissue disorders) | 0 | 4
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 3 | 5
PHLEBITIS (Vascular disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.